CLINICAL TRIAL: NCT00006011
Title: A Randomized Phase III Study of Tumor Volume Directed Pelvic Plus or Minus Para-Aortic Irradiation Followed by Cisplatin and Doxorubicin or Cisplatin, Doxorubicin and Paclitaxel for Advanced Endometrial Carcinoma
Brief Title: Comparison of Two Combination Chemotherapy Regimens Plus Radiation Therapy in Treating Patients With Stage III or Stage IV Endometrial Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: Eastern Cooperative Oncology Group (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GOG-0184; NCI-2012-02350 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-G0184; RTOG-EN0130; CDR0000068020; GOG-0184 (Other: Gynecologic Oncology Group); GOG-0184 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-04

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Adenosquamous Carcinoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Endometrioid Adenocarcinoma, Variant With Squamous Differentiation; Endometrial Serous Adenocarcinoma; Stage III Uterine Corpus Cancer
MeSH Terms: interventions — Doxorubicin; Cisplatin; Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim; Paclitaxel; Taxes

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (doxorubicin, cisplatin, filgrastim, pegfilgrastim) (Experimental): Patients receive doxorubicin IV over 30 minutes immediately followed by cisplatin IV over 1 hour on day 1. Patients also receive filgrastim (G-CSF) SC or pegfilgrastim on days 2-11.
  Interventions: Drug: Doxorubicin Hydrochloride; Drug: Cisplatin; Biological: Filgrastim; Biological: Pegfilgrastim
- Arm II (doxorubicin, cisplatin, paclitaxel, filgrastim) (Experimental): Patients receive doxorubicin and cisplatin as in arm I, paclitaxel IV over 3 hours on day 2, and G-CSF SC or pegfilgrastim on days 3-12. Treatment repeats every 3 weeks for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Doxorubicin Hydrochloride; Drug: Cisplatin; Biological: Filgrastim; Biological: Pegfilgrastim; Drug: Paclitaxel

INTERVENTIONS:
Drug: Doxorubicin Hydrochloride — Given IV
Drug: Cisplatin — Given IV
Biological: Filgrastim — Given SC
  Other Names: G-CSF; Nivestim; r-metHuG-CSF
Biological: Pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; GCSF-SD01; Neulasta
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; TAX
  Arms: Arm II (doxorubicin, cisplatin, paclitaxel, filgrastim)

SUMMARY:
Randomized phase III trial to compare the effectiveness of two combination chemotherapy regimens plus radiation therapy in treating patients who have stage III or stage IV endometrial cancer. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one chemotherapy drug with radiation therapy may kill more tumor cells. It is not yet known which combination chemotherapy regimen plus radiation therapy is more effective for endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare survival and progression-free survival in patients with stage III endometrial carcinoma treated with tumor volume-directed pelvic radiotherapy with or without paraaortic radiotherapy followed by cisplatin and doxorubicin with or without paclitaxel.

II. Compare short and long-term toxic effects of these treatment regimens in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to radiotherapy field (pelvic vs extended field). Within 8 weeks after surgery, patients receive tumor volume-directed pelvic radiotherapy with or without paraaortic nodal radiotherapy once daily for 5 consecutive days for up to 16 weeks after surgery. Within 8 weeks of completing radiotherapy, patients are randomized to 1 of 2 chemotherapy treatment arms.

Arm I: Patients receive doxorubicin IV over 30 minutes immediately followed by cisplatin IV over 1 hour on day 1. Patients also receive filgrastim (G-CSF) subcutaneously (SC) or pegfilgrastim on days 2-11.

Arm II: Patients receive doxorubicin and cisplatin as in arm I, paclitaxel IV over 3 hours on day 2, and G-CSF SC or pegfilgrastim on days 3-12. Treatment repeats every 3 weeks for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 614 patients (307 per treatment arm) will be accrued for this study within 5.2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced endometrial carcinoma with any histology, including:

  * Clear cell and serous papillary carcinoma
* Surgical stage III disease, including:

  * Positive adnexa
  * Tumor invading the serosa
  * Positive pelvic and/or paraaortic nodes
  * Involvement of bowel mucosa
  * Intraabdominal metastases
  * Positive pelvic washings
  * Vaginal involvement within the radiation port
* Must have had prior surgery, including hysterectomy and bilateral salpingo-oophorectomy

  * Tumor maximally debulked to a maximum residual diameter of no greater than 2 cm
  * Paraaortic lymph node sampling allowed

    * If positive, must have negative chest CT scan
* No recurrent disease
* No parenchymal liver metastases
* No disease outside the abdomen
* Performance status - GOG 0-2
* At least 3 months
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times normal
* SGOT/SGPT no greater than 3 times normal
* Alkaline phosphatase no greater than 3 times normal
* Creatinine no greater than 1.6 mg/dL
* LVEF at least 50% within 6 months of study entry
* No other prior or concurrent malignancy within the past 5 years except adequately treated nonmelanoma skin cancer
* No serious comorbid illness that would preclude study participation
* No prior chemotherapy
* See Disease Characteristics
* No prior pelvic or abdominal radiotherapy
* No prior radiotherapy for prior malignancy
* See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 659 (Actual)
Dates: Start 2000-07; Primary Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Homesley, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were initially registered and initiated radiation treatment. Following succsessful completion of radiation treatment, participants with no evidence of disease received a random treatment allocation.
Groups:
- Arm 1: Treatment randomization following RT.
  radiation followed by doxorubicin 45 mg/m2 and cisplatin 50 mg/m2 G-CSF 5mcg/kg Days 2-11
- Arm 2: Treatment randomization following RT:
  radiation followed by doxorubicin 45 mg/m2 and cisplatin 50 mg/m2 day 1 paclitaxel 3-Hr 160 mg/m2 day 2 G-CSF 5 mcg/kg days 3-12
- Radiation (RT) Only: Tumor volume directed pelvic plus or minus para-aortic irradiation (plus or minus brachytherapy)
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Radiation (RT) Only
Started | 288 (total number of participants enrolled, that received random treatment assignment to Arm 1 of study.) | 298 (total number of participants enrolled, that received random treatment assignment to Arm 2 of study.) | 73 (total number of participants enrolled, that only received radiation treatment.)
Completed | 223 (total number of partipants that completed 6 cycles of chemotherapy.) | 221 (total number of partipants that completed 6 cycles of chemotherapy.) | 0 (total number of partipants that completed 6 cycles of chemotherapy.)
Not Completed | 65 | 77 | 73
Not completed — Disease progression | 13 | 6 | 26
Not completed — Refused further treatment | 15 | 13 | 26
Not completed — Adverse Event | 15 | 39 | 5
Not completed — Death | 0 | 1 | 2
Not completed — Other | 4 | 2 | 5
Not completed — Ineligible | 18 | 16 | 9

BASELINE CHARACTERISTICS:
Population: Total number of eligible participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Radiation (RT) Only | Total
Number analyzed (Participants) | 270 | 282 | 64 | 616
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (11.1) | 58.8 (9.5) | 63.9 (10.7) | 59.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 270 | 282 | 64 | 616
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-Free Survival of Eligible Patients Who Received a Random Treatment Allocation.
Description: Recurrence is defined as discovery of disease not previously present by clinical, radiographic, and/or laboratory means or as a 50% or greater increase in the product of two perpendicular diameters from any documented lesion.
  Recurrence-free survival is defined as time in months the patient is alive, recurrence-free starting from the date of randomization.
  Intention to treat among eligible participants who receive random treatment allocation.
Time Frame: study entry up to 5 years post treatment
Measure: Number; unit: participants
Groups:
- Arm 1: Treatment randomization following RT.
  doxorubicin 45 mg/m2 and cisplatin 50 mg/m2 G-CSF 5mcg/kg Days 2-11
- Arm 2: Treatment randomization following RT:
  doxorubicin 45 mg/m2 and cisplatin 50 mg/m2 day 1 paclitaxel 3-Hr 160 mg/m2 day 2 G-CSF 5 mcg/kg days 3-12
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 270 | 282
participants
  Alive, Recurrence-Free | 159 | 175
  Recurrence or Death | 111 | 107
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Primary outcome is measured as a treatment hazard ratio stratified by stage and assuming proportional hazards. Recurrence-free survival hazard ratio: Arm 2 is relative to Arm 1; Test type: Superiority or Other; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.69 to 1.17]

ADVERSE EVENTS:
Time Frame: The frequencies of any serious adverse event or other adverse events by category or specific term occurring during chemotherapy treatment and up to 30 days after stopping the study treatment are reported.
Description: Serious Adverse Events(SAE) are reported separately. Due to the methods in which AEs were collected &/or stored, it isn't possible to report Other AEs separate from SAEs. That table is a combined set of SAEs & non-serious AEs. Other AEs are acute, grade 2 or worse AEs that occured during chemotherapy treatmentand don't include late AEs.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 10/261 | 21/278
Other Adverse Events (participants affected / at risk) | 259/261 | 278/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=261) | Arm 2 (N=278)
Dehydration (Gastrointestinal disorders) | 0 | 1
Cns Cerebrovascular Ischemia (Nervous system disorders) | 1 | 1
Neutrophils/Granulocytes (Blood and lymphatic system disorders) | 0 | 3
Circulatory or Cardia, Other (Cardiac disorders) | 0 | 1
Hypotension (Cardiac disorders) | 0 | 1
Vasovagal Episode (Cardiac disorders) | 0 | 1
Supraventricular Arrhythmias (Cardiac disorders) | 0 | 2
Cardia-Ischemia/Infarction (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Abdominal Pain or Cramping (General disorders) | 1 | 1
Pain, Other (General disorders) | 0 | 1
Wound-Infectious (Skin and subcutaneous tissue disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Anorexia (Gastrointestinal disorders) | 1 | 0
Diarrhea (without Colostomy) (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1
Infection, Other (Infections and infestations) | 1 | 0
Infection Documented with Grade 3/4 Neutropenia (Infections and infestations) | 0 | 1
Infection without Neutropenia (Infections and infestations) | 1 | 0
Febrile Neutropenia-Fuo Infection Not Documented (Infections and infestations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Osteonecrosis (Avascular Necrosis) (Musculoskeletal and connective tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Neuropathy-Sensory (Nervous system disorders) | 0 | 1
Thrombosis/Embolism (Vascular disorders) | 0 | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=261) | Arm 2 (N=278)
Leukopenia (Blood and lymphatic system disorders) | 190 | 250
Neutropenia (Blood and lymphatic system disorders) | 158 | 236
Thrombocytopenia (Blood and lymphatic system disorders) | 55 | 116
Anemia (Blood and lymphatic system disorders) | 137 | 205
Other Hematologic (Blood and lymphatic system disorders) | 44 | 71
Allergy (Immune system disorders) | 4 | 8
Auditory (Ear and labyrinth disorders) | 16 | 8
Cardiac left ventricular function (Cardiac disorders) | 28 | 24
Other Cardiovascular (Cardiac disorders) | 29 | 44
Coagulation (Cardiac disorders) | 0 | 4
Constitutional (General disorders) | 105 | 133
Alopecia (Skin and subcutaneous tissue disorders) | 185 | 179
Other Dermatologic (Skin and subcutaneous tissue disorders) | 15 | 17
Endocrine (Endocrine disorders) | 17 | 14
Nausea (Gastrointestinal disorders) | 89 | 95
Vomiting (Gastrointestinal disorders) | 75 | 79
Stomatitis (Gastrointestinal disorders) | 11 | 15
Other Gastrointestinal (Gastrointestinal disorders) | 73 | 88
Genitourinary/Renal (Renal and urinary disorders) | 18 | 27
Hemorrhage (Vascular disorders) | 2 | 5
Hepatic (Renal and urinary disorders) | 6 | 14
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 17
Infection Without Neutropenia (Infections and infestations) | 25 | 32
Other Infection/Fever (Infections and infestations) | 11 | 35
Lymphatics (Blood and lymphatic system disorders) | 5 | 5
Metabolic (Metabolism and nutrition disorders) | 46 | 55
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 11 | 26
Peripheral Sensory Neurologic (Nervous system disorders) | 13 | 76
Other Neurologic (Nervous system disorders) | 31 | 52
Ocular/Visual (Eye disorders) | 11 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 52
Other Pain (General disorders) | 63 | 101
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 31 | 39
Sexual (Reproductive system and breast disorders) | 3 | 5
2nd Primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 18 — 2nd primary is not necessarily secondary malignancy and may have been reported any time after randomization including the follow-up period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No